CLINICAL TRIAL: NCT06149702
Title: A Feasibility Randomised Controlled Trial of a Digital Program to Prevent Falls and Improve Well-being in People Living With Dementia in the Community.
Brief Title: A Digital Health App to Prevent Falls and Improve Well-being in People Living With Dementia
Acronym: KOKU-D
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jaheeda Gangannagaripalli (Other)
Responsible Party: Sponsor-Investigator, Jaheeda Gangannagaripalli, Dr, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Version 3.1, 13.05.24
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Dementia
Keywords: Quality of life; Well-being; Dementia; Feasibility study; Technology; Falls prevention; strength and balance
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This feasibility randomised controlled trial is a 6-week study comparing the intervention (KOKU-LITE programme + dementia and falls prevention leaflet) to control (dementia and falls prevention leaflet) in community dwelling people living with dementia and carers of people living with dementia. After assessing participants for eligibility, they will be allocated randomly to either intervention group or control group. Assessments will be performed at baseline and 6 weeks post follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Keep-on-Keep-Up-LITE (KOKU-LITE) programme and dementia and falls prevention leaflet (Other): Intervention arm: Keep-on-Keep-Up-LITE (KOKU-LITE) programme and dementia and falls prevention leaflet.
  Participants will attend a KOKU-LITE training session lasting for 60 minutes. A carer may also accompany if the participant feels that their support would be beneficial. An iPad will be provided to participants for the duration of the project and the app instruction booklet will also be provided for reference purposes. For participants who do not wish to attend the group training, ad hoc one-to-one training will be offered. * Participants will be advised to use KOKU-LITE for 30 minutes, 3 times per week, for 6 weeks and also read the dementia and falls prevention leaflet
  Interventions: Other: Combined intervention: Keep-on-Keep-Up-LITE (KOKU-LITE) programme and dementia and falls prevention leaflet
- Control arm (Dementia and Falls prevention leaflet) (Other): If participants are allocated to the intervention group, they will use KOKU-LITE for 30 minutes 3 times a week for 6 weeks along with the dementia and falls prevention leaflet. If participants are allocated to the control group, they will receive Dementia and Falls prevention leaflet (https://www.dementiauk.org/wp-content/uploads/dementia-uk-falls.pdf)l (and not use KOKU-LITE).
  Interventions: Other: Combined intervention: Keep-on-Keep-Up-LITE (KOKU-LITE) programme and dementia and falls prevention leaflet

INTERVENTIONS:
Other: Combined intervention: Keep-on-Keep-Up-LITE (KOKU-LITE) programme and dementia and falls prevention leaflet — KOKU-LITE programme will be used by the participants for 6 weeks and outcome assessments will be performed at baseline and 6 weeks of use. Participants will also use dementia and falls prevention leaflet for 6 weeks.

SUMMARY:
"Keep on Keep up (KOKU)" is a tablet/iPad-based, digital strength and balance exercise programme specifically designed for older people at risk of falls. Research has shown that the exercises reduce falls by around a third in older people. People with Dementia are more reluctant and have greater challenges with using digital technologies. Evidence suggests that developing technologies in a Patient-Centered manner will be more acceptable in this population as People living with Dementia are more reluctant to using digital technologies. The existing version of the KOKU digital programme has been modified in collaboration with People living with Dementia and carers of People living with Dementia to suit their needs and make it Dementia-friendly, and accessible to People living with Dementia known as KOKU-LITE. The current project involves testing KOKU-LITE with People living with Dementia, their carers, and health and social care professionals. This project will have many possible benefits for People living with Dementia; It has the potential to improve quality of life (QoL), well-being, confidence, independence, and therefore has the potential to reduce general practice visits, hospital admissions, and health and social care costs.

ELIGIBILITY:
Inclusion Criteria:

Participant inclusion criteria:

People living with dementia (PLwD) and carers of PLwD Participants will be selected purposively to derive a maximum variation sample including age, gender, diverse representation from different backgrounds and different levels of Dementia, early cognitive decline and different stages of disease progression thus, increase the external generalisability of the results.

* PLwD and carers of PLwD aged ≥55 yrs
* willing and able to give informed consent (assessed by the trained researchers and/or health and social care professionals (HSCPs)).
* who lack capacity to consent themselves but can be supported by a carer or an advocate.
* Carers of PLwD who lack capacity to consent themselves.
* able to speak English.
* able to see the tablet/iPad-based app and read instructions with or without glasses.
* able to use tablet/iPad safely, as assessed by the trained research staff and/or HSCPs.
* able to move indoors without help, and with or without a walking aid.

Professionals

• HSCPs caring for PLwD

Exclusion Criteria:

PLwD

* Participants with:

  * Acute/chronic or uncontrolled medical condition (e.g. severe congestive cardiac failure, uncontrolled hypertension, acute systemic illness, neurological problems, poorly controlled diabetes).
  * recent fracture or surgery (within 6 months)
  * orthopaedic surgery (such as hip/knee surgery) in the past six months or on a waiting list to have the surgery.
  * heart problems such as myocardial infarction or stroke in the past six months
  * conditions requiring a specialist/exercise programme (e.g., uncontrolled epilepsy, or uses a wheelchair to mobilise indoors).
  * severe hearing/visual impairment.
  * any other medical condition likely to compromise the ability to use/access the app.
* Participants currently in hospital or care home,
* Participants who have limited understanding or ability to speak English, and .
* Persons with Dementia who do not have a carer who can provide assent.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The feasibility and acceptability of the intervention | 6 weeks
  The feasibility and acceptability of the intervention will be evaluated in terms of recruitment, retention and adherence rates to the trial. This will be evaluated by calculating the percentage of people approached who participate in the trial (recruitment) and the percentage of participants who complete the trial (including using KOKU-LITE and dementia and falls prevention leaflet and completing the questionnaires) (retention and adherence).

SECONDARY OUTCOMES:
Health-related Quality of life will be measured using EQ-5D-5L scale | 6 weeks: Health-related Quality of life will measured at baseline and 6 weeks post follow-up
  Health-related Quality of life as measured by The European Quality of Life 5 Dimensions (EQ-5D-5L) scale.
  EQ-5D-5L is a 5-dimension version of the original EQ-5D scale. It has two sections: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The 5 responses give a health state or profile represented by a 5-digit number (for example, 12231) corresponding to response categories reported by patients for successive dimensions: mobility, self care, usual activities, pain/discomfort, anxiety/depression. Current recommendations for scoring the EQ-5D-5L index will be followed. Index scores range from -0.59 to 1; 1 is the best possible health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where 0 indicates 'worst health you can imagine' and 100 indicates 'the best health you can imagine'.
The Erlangen Test for Activities of Daily Living test | 6 weeks: E-ADL-Test will be assessed at baseline and 6 weeks post-follow up
  The Erlangen Test for Activities of Daily Living test (E-ADL-Test) is a valid and reliable instrument for assessing the ADL capabilities of people with Dementia. It includes 4 domains: Pouring a drink, Cutting a piece of bread, Opening a little cupboard, Washing hands.
  The total score of the E-ADL ranges from 0-30, with a higher score representing better results.
Short Physical Performance Battery | 6 weeks: participants will be assessed at baseline and 6 weeks post-follow up using SPPB
  The Short Physical Performance Battery (SPPB) is a validated and reliable instrument to assess functional mobility in people with cognitive impairment/dementia. SPPB is a validated and reliable instrument to assess functional mobility in people with cognitive impairment/dementia. The SPPB test includes three different domains: walking, sit-to-stand and balance. The scores range from 0 (worst performance) to 12 (best performance).
Geriatric Depression Scale | 6 weeks: The 5-item Geriatric Depression Scale screening tool will be measured at baseline and 6 weeks post follow-up
  The 5-item Geriatric Depression Scale screening tool for depression in older adults. The 5-item Geriatric Depression Scale screening tool for depression in older adults (validated to be as effective as the 15-item GDS for older adults in a wide range of settings). A score of 0 to 1 for the 5-item GDS suggests that the subject is not depressed, while 2 or higher indicates possible depression.
Falls risk will be measured with the use of the Assessment of falls risk tool. | 6 weeks: FRAT tool will be measured at baseline and 6 weeks post follow-up
  Falls risk will be measured with the use of the Assessment of falls risk (FRAT) tool. (VI) Falls risk will be measured with the use of the Assessment of falls risk (FRAT) tool. This validated measure has 5 items which include; history of any fall in the previous year, four or more prescribed medications, diagnosis of stroke or Parkinson's disease, reported problems with balance and inability to rise from a chair without using arms. These are all strong indicators for risk of falling. If a person scores 3 or more they are at high risk of falling.
Short Falls Efficacy Scale-International | 6 weeks: FES-1 scale will be measured at baseline and 6 weeks post-follow up
  The Short Falls Efficacy Scale-International (FES-I). The FES-I is a validated and reliable 7-item tool that measures confidence in performing a range of activities of daily living without falling. This scale has recently been modified to maximise its suitability for a range of different languages and cultures. Scoring: Minimum 7 (no concern about falling) to maximum 28 (severe concern about falling).
The User Experience Questionnaire | UEQ will only be measured at 6 weeks post-follow up in the intervention group only (to those who use KOKU-LITE))
  The User Experience Questionnaire (UEQ) is a standardized 26-item questionnaire that is used reliably to assess the quality and user experience of the interactive products. The standard interpretation of the scale means is that values between -0.8 and 0.8 represent a neural evaluation of the corresponding scale, values > 0,8 represent a positive evaluation and values < -0,8 represent a negative evaluation. The range of the scales is between -3 (horribly bad) and +3 (extremely good).

CONTACTS AND LOCATIONS:
Overall Officials: Jaheeda Begum Gangannagaripalli, PhD, Principal Investigator — The University of Manchester
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At the end of the project, we will deposit a fully anonymised dataset [including de-identified interview transcripts] in an open data repository where it will be permanently stored. We will use Figshare at the University of Manchester Library. Researchers at other institutions and others can access the anonymised data directly from the repository and use it for further research or to check our analysis and results.

REFERENCES:
- [Derived] Gangannagaripalli J, Vardy E, Stanmore E. A digital programme to prevent falls and improve well-being in people living with dementia in the community: the KOKU-LITE feasibility randomised controlled trial protocol. BMJ Open. 2025 Aug 19;15(8):e091222. doi: 10.1136/bmjopen-2024-091222. PMID 40829848